CLINICAL TRIAL: NCT03347435
Title: Pharmacogenetics of Clopidogrel in Acute Coronary Syndromes
Acronym: PHARMCLO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Ethics Committe decision
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Diego Ardissino, Director of Division of Cardiology, Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11210
Record Dates: First submitted 2017-11-10; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Acute Coronary Syndromes
Keywords: clopidogrel; pharmacogenetics; antiplatelet therapy; acute coronary syndromes
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Genotype/ phenotype guided group (Experimental): The patients randomized to the genotype/phenotype guided group undergo genetic tests for CYP2C19*2, CYP2C19*17 and ABCB1 3435 genetic variants immediately after diagnosis of ACS and receive one of the ADP receptor antagonists (clopidogrel/prasugrel/ticagrelor) on the basis of an algorithm that consider genetic and clinical variables.
  Interventions: Genetic: genetic tests for CYP2C19*2, CYP2C19*17 and ABCB1 3435
- phenotype only guided group (Active Comparator): The patients randomized to the phenotype only guided group receive clopidogrel or prasugrel or ticagrelor on the basis of the standard of care on the basis of clinical algorithm alone.
  Interventions: Other: clinical algorithm

INTERVENTIONS:
Genetic: genetic tests for CYP2C19*2, CYP2C19*17 and ABCB1 3435 — The CYP2C19*2 (10q24.1-q24.3; rs4244285), CYP2C19*17 (10q24.1-q24.3; rs12248560) and ABCB1 3435 (7q21.1; rs1045642) genetic variants will be genotyped using an ST Q3 system. The conventional genotyping methods so far used for diagnostic purposes will not be used in this study because appropriate labs may not be readily available and the processing time is prohibitive. Q3 is a compact platform enabling the classical laboratory analysis of DNA by means of real-time PCR. The Q3 has been designed as a low entry-cost, portable, point-of-care instrument for foolproof use by unskilled personnel. Antiplatelet therapy will be choose on the basis of clinical and genetic algorithm.
  Arms: Genotype/ phenotype guided group
Other: clinical algorithm — Antiplatelet therapy will be choose on the basis of clinical algorithm alone
  Arms: phenotype only guided group

SUMMARY:
The antiplatelet agent clopidogrel is an effective drug for the prevention of thrombotic events in patients with acute coronary syndromes, and is therefore one of the most frequently prescribed drugs worldwide. Accumulating data suggest that the response to clopidogrel is characterised by significant inter-patient variability in the degree of platelet inhibition and the risk of cardiovascular events. Recent research findings have highlighted the role of genetic variations in determining antiplatelet response variability, and this has aroused interest in genotyping all thienopyridine-eligible patients in order to identify those who would be at increased risk of harm if treated with clopidogrel. This is a prospective, multicentre, randomised study enrolling consecutive patients hospitalised because of an ACS with or without ST-segment elevation. The patients are randomised to undergo or not tests for CYP2C19*2, CYP2C19*17 and ABCB1 3435 genetic variants immediately after diagnosis. The genotyping is done using a Q3 System (a compact platform that enables the classic laboratory analysis of DNA by means of real-time PCR). The Q3 has been designed as a low entry-cost, portable, point-of-care instrument for foolproof use by unskilled personnel. The patients randomised to the pharmacogenomic arm receive one of the ADP receptor antagonists (clopidogrel/prasugrel/ticagrelor) on the basis of an algorithm that consider genetic and clinical variables. The patients randomised to the standard treatment arm receive clopidogrel or prasugrel or ticagrelor on the basis of the standard of care (clinical algorithm alone). For each patient, a record is made of the occurrence of cardiovascular death, non-fatal MI, stroke, BARC-defined bleeding, and definite or probable stent thrombosis. The primary endpoint is the composite of death due to cardiovascular causes, non-fatal MI and stroke. The secondary endpoints is the occurrence of definite or probable stent thrombosis, and BARC-defined major bleeding events (types 3-5).

DETAILED DESCRIPTION:
Antiplatelet therapy is the cornerstone of medical treatment of patients experiencing an acute coronary syndrome (ACS). As a synergistic antiplatelet effect can be obtained by simultaneously inhibiting thromboxane-A2 and adenosine diphosphate P2Y12 platelet receptors, the current standard of care for all patients with ACS includes dual anti-platelet therapy with aspirin (the first choice treatment for blocking thromboxane-A2 receptors) and one of the three currently available ADP P2Y12 inhibitors: clopidogrel, prasugrel and ticagrelor.

Over the last few years, the clinical availability of the new potent P2Y12 inhibitors prasugrel and ticagrelor has changed the ACS treatment paradigm. The revised European guidelines downgrade clopidogrel to patients who cannot receive prasugrel and ticagrelor, and clearly recommend the latter for patients with ACS (Recommendation Class I, Evidence Level B for both). However, the choice of the optimal drug for each individual patient is still left to clinicians, thus continuing the uncertainty as to how these new potent drugs should be incorporated into everyday clinical practice.

The appropriate selection of antiplatelet agents has so far been guided only by the patients' phenotypic characteristics, but taken together, the evidence does not support a wide use of prasugrel and ticagrelor in clinical practice and considering subgroups with less clinical benefit and limitations of TRITON TIMI-38 and PLATO study design, not all 100% of patients with ACS appears eligible for treatment with new ADP receptors antagonists.

Recent research has highlighted the role of CYP enzyme and ABCB1 genetic variations in determining the variability of the patients' antiplatelet response to clopidogrel, and shown a clear relationship between lower levels of clopidogrel's active metabolite, reduced platelet inhibition, and a higher rate of major adverse cardiovascular events. Specifically, post-hoc analysis concerning association of CYP2C19 and ABCB1 genetic variants to clinical outcomes showed an absolute 7.3% reduction in the risk of death from cardiovascular causes, myocardial infarction or stroke among the study population who were not carriers of a CYP2C19 reduced-function allele, ABCB1 3435 TT homozygotes, or both, compared with individuals who did carry either.

The impact of CYP2C19 alleles and ABCB1 genotype seems to be restricted to patients taking clopidogrel as they do not significantly affect pharmacological or clinical outcomes in patients treated with prasugrel and ticagrelor.

The aim of this project is to test the impact on clinical outcomes of strategy of conducting dual antiplatelet therapy considering both genotype data and clinical variables in comparison with a strategy based on clinical variables alone.

Methodology:

This is a prospective, multicentre, randomised study enrolling 3,612 consecutive patients hospitalised because of an ACS with or without ST-segment elevation. The patients are randomised to undergo or not tests for CYP2C19*2, CYP2C19*17 and ABCB1 3435 genetic variants immediately after diagnosis. The genotyping is done using a Q3 System (a compact platform that enables the classic laboratory analysis of DNA by means of real-time PCR). The Q3 has been designed as a low entry-cost, portable, point-of-care instrument for foolproof use by unskilled personnel.

The patients randomised to the pharmacogenomic arm receive one of the ADP receptor antagonists (clopidogrel/prasugrel/ticagrelor) on the basis of an algorithm that consider genetic and clinical variables. The patients randomised to the standard treatment arm receive clopidogrel or prasugrel or ticagrelor on the basis of the standard of care (clinical algorithm alone).

Patient enrolment is to be completed in 24 months. Each patient will be followed up for 12 months by means of outpatient visits after one, six and 12 months.

For each patient, a record is made of the occurrence of cardiovascular death, non-fatal MI, stroke, BARC-defined bleeding, and definite or probable stent thrombosis.

The primary endpoint is the composite of death due to cardiovascular causes, non-fatal MI and stroke.

The secondary endpoints is the occurrence of definite or probable stent thrombosis, and BARC-defined major bleeding events (types 3-5).

The expected rate reduction of ischemic and bleeding events is 25% for a median of 12 months of follow-up (data derived from PLATO trial) and the target relative risk reduction for genotype-guided therapy versus standard therapy is 20%. It has been defined a 95% power, a type alpha error of 5% and two-tail test. Therefore approximately 1806 patients for each arm should be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ACS (STE-ACS or NSTE-ACS) during the index hospitalisation
* Age >18 years
* Ability to sign the informed consent form
* Ability to attend scheduled visits

Exclusion Criteria:

* Cognitive or other causes of an inability to provide informed consent or follow study procedures
* Any contraindication to the use of ADP P2Y12 inhibitors
* Life expectancy <1 year
* Thrombolytic therapy within the previous 24 hours
* Known ABCB1, CYP2C19 *2 orCYP2C19 *17 genotype

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 889 (Actual)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Composite of cardiovascular death, non fatal myocardial infarction, stroke and BARC-defined major bleeding events 3 to 5. | 12 months
  The primary endpoint will be the composite of cardiovascular death, non fatal myocardial infarction, stroke and BARC-defined major bleeding events 3 to 5 at 12 months follow-up.

SECONDARY OUTCOMES:
occurrence of definite or probable stent thrombosis. | 12 months
  The secondary endpoint variable will be the occurrence of definite or probable stent thrombosis at 12 months follow-up.
cardiovascular death | 12 months
  individual components of primary endpoint at 12 months follow-up
non fatal myocardial infarction | 12 months
  individual components of primary endpoint at 12 months follow-up
stroke | 12 months
  individual components of primary endpoint at 12 months follow-up
BARC-defined major bleeding events 3 to 5 | 12 months
  individual components of primary endpoint at 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Diego Ardissino, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma
Locations (4):
- Italy (4):
  - Ospedale Ramazzini, Carpi, Modena
  - Ospedale di Vaio, Fidenza, Parma
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Ospedale Guglielmo da Saliceto, Piacenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hamm CW, Bassand JP, Agewall S, Bax J, Boersma E, Bueno H, Caso P, Dudek D, Gielen S, Huber K, Ohman M, Petrie MC, Sonntag F, Uva MS, Storey RF, Wijns W, Zahger D; ESC Committee for Practice Guidelines. ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: The Task Force for the management of acute coronary syndromes (ACS) in patients presenting without persistent ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2011 Dec;32(23):2999-3054. doi: 10.1093/eurheartj/ehr236. Epub 2011 Aug 26. No abstract available. PMID 21873419
- [Result] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Result] Wiviott SD, Braunwald E, McCabe CH, Montalescot G, Ruzyllo W, Gottlieb S, Neumann FJ, Ardissino D, De Servi S, Murphy SA, Riesmeyer J, Weerakkody G, Gibson CM, Antman EM; TRITON-TIMI 38 Investigators. Prasugrel versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2007 Nov 15;357(20):2001-15. doi: 10.1056/NEJMoa0706482. Epub 2007 Nov 4. PMID 17982182
- [Result] Matetzky S, Shenkman B, Guetta V, Shechter M, Beinart R, Goldenberg I, Novikov I, Pres H, Savion N, Varon D, Hod H. Clopidogrel resistance is associated with increased risk of recurrent atherothrombotic events in patients with acute myocardial infarction. Circulation. 2004 Jun 29;109(25):3171-5. doi: 10.1161/01.CIR.0000130846.46168.03. Epub 2004 Jun 7. PMID 15184279
- [Result] Mega JL, Close SL, Wiviott SD, Shen L, Hockett RD, Brandt JT, Walker JR, Antman EM, Macias W, Braunwald E, Sabatine MS. Cytochrome p-450 polymorphisms and response to clopidogrel. N Engl J Med. 2009 Jan 22;360(4):354-62. doi: 10.1056/NEJMoa0809171. Epub 2008 Dec 22. PMID 19106084
- [Result] Shuldiner AR, O'Connell JR, Bliden KP, Gandhi A, Ryan K, Horenstein RB, Damcott CM, Pakyz R, Tantry US, Gibson Q, Pollin TI, Post W, Parsa A, Mitchell BD, Faraday N, Herzog W, Gurbel PA. Association of cytochrome P450 2C19 genotype with the antiplatelet effect and clinical efficacy of clopidogrel therapy. JAMA. 2009 Aug 26;302(8):849-57. doi: 10.1001/jama.2009.1232. PMID 19706858
- [Result] Mega JL, Close SL, Wiviott SD, Shen L, Walker JR, Simon T, Antman EM, Braunwald E, Sabatine MS. Genetic variants in ABCB1 and CYP2C19 and cardiovascular outcomes after treatment with clopidogrel and prasugrel in the TRITON-TIMI 38 trial: a pharmacogenetic analysis. Lancet. 2010 Oct 16;376(9749):1312-9. doi: 10.1016/S0140-6736(10)61273-1. PMID 20801494
- [Result] Wallentin L, James S, Storey RF, Armstrong M, Barratt BJ, Horrow J, Husted S, Katus H, Steg PG, Shah SH, Becker RC; PLATO investigators. Effect of CYP2C19 and ABCB1 single nucleotide polymorphisms on outcomes of treatment with ticagrelor versus clopidogrel for acute coronary syndromes: a genetic substudy of the PLATO trial. Lancet. 2010 Oct 16;376(9749):1320-8. doi: 10.1016/S0140-6736(10)61274-3. PMID 20801498
- [Result] Tiroch KA, Sibbing D, Koch W, Roosen-Runge T, Mehilli J, Schomig A, Kastrati A. Protective effect of the CYP2C19 *17 polymorphism with increased activation of clopidogrel on cardiovascular events. Am Heart J. 2010 Sep;160(3):506-12. doi: 10.1016/j.ahj.2010.06.039. PMID 20826260
- [Result] Mega JL, Simon T, Collet JP, Anderson JL, Antman EM, Bliden K, Cannon CP, Danchin N, Giusti B, Gurbel P, Horne BD, Hulot JS, Kastrati A, Montalescot G, Neumann FJ, Shen L, Sibbing D, Steg PG, Trenk D, Wiviott SD, Sabatine MS. Reduced-function CYP2C19 genotype and risk of adverse clinical outcomes among patients treated with clopidogrel predominantly for PCI: a meta-analysis. JAMA. 2010 Oct 27;304(16):1821-30. doi: 10.1001/jama.2010.1543. PMID 20978260
- [Result] Sibbing D, Koch W, Gebhard D, Schuster T, Braun S, Stegherr J, Morath T, Schomig A, von Beckerath N, Kastrati A. Cytochrome 2C19*17 allelic variant, platelet aggregation, bleeding events, and stent thrombosis in clopidogrel-treated patients with coronary stent placement. Circulation. 2010 Feb 2;121(4):512-8. doi: 10.1161/CIRCULATIONAHA.109.885194. Epub 2010 Jan 18. PMID 20083681
- [Derived] Notarangelo FM, Maglietta G, Bevilacqua P, Cereda M, Merlini PA, Villani GQ, Moruzzi P, Patrizi G, Malagoli Tagliazucchi G, Crocamo A, Guidorossi A, Pigazzani F, Nicosia E, Paoli G, Bianchessi M, Comelli MA, Caminiti C, Ardissino D. Pharmacogenomic Approach to Selecting Antiplatelet Therapy in Patients With Acute Coronary Syndromes: The PHARMCLO Trial. J Am Coll Cardiol. 2018 May 1;71(17):1869-1877. doi: 10.1016/j.jacc.2018.02.029. Epub 2018 Mar 11. PMID 29540324